CLINICAL TRIAL: NCT00515632
Title: A Randomized, Double-blind, Parallel-group, Placebo and Active Comparator (Pioglitazone)-Controlled Clinical Study to Determine the Efficacy and Safety of Balaglitazone in Patients With Type 2 Diabetes on Stable Insulin Therapy
Brief Title: Efficacy and Safety of Treatment With Balaglitazone in Type 2 Diabetes Patients on Stable Insulin Therapy
Acronym: BALLET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rheoscience A/S (Other)
Responsible Party: Bente Juel Riis, MD, Rheoscience A/S
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRF2593-307; EudraCT No. 2007-002088-29
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes mellitus on Stable insulin therapy; Balaglitazone; Pioglitazone (Actos®); HbA1c; Weight gain; Oedema; Fasting blood glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Weight Gain; Edema | interventions — balaglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Balaglitazone 10 mg per day (Experimental)
  Interventions: Drug: Balaglitazone
- Balaglitazone 20 mg per day (Experimental)
  Interventions: Drug: Balaglitazone
- Pioglitazone 45 mg per day (Active Comparator)
  Interventions: Drug: Balaglitazone
- Placebo (Placebo Comparator)
  Interventions: Drug: Balaglitazone

INTERVENTIONS:
Drug: Balaglitazone — One arm balaglitazone 10mg, one arm balaglitazone 20mg, one arm placebo, one arm pioglitazone (Actos®) 45mg, orally taken once daily.

SUMMARY:
Type 2 diabetes mellitus is a metabolic disorder that is primarily characterized by insulin resistance, relative insulin deficiency, and hyperglycemia. People with type 2 diabetes are at high risk of many serious diabetic complications, including cardiovascular disease, blindness, nerve damage and kidney damage. Balaglitazone is a thiazolidinedione derivative that is being developed as an oral anti-diabetic drug to improve blood glucose control in patients with type 2 diabetes. The purpose of this study is to assess if additional treatment with balaglitazone in patients with type 2 diabetes on stable insulin treatment will improve blood glucose control and decrease the daily insulin dose compared to placebo, but with less impact on weight gain and oedema than pioglitazone (Actos®) 45 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus, being diagnosed according to the 1999 WHO criteria for at least 3 months
2. Age ≥ 18 years
3. BMI ≥ 25.0 kg/m2
4. HbA1c ≥ 7.0 %
5. Treatment with insulin with stable dose of at least 30 U/day (± 4 U/day), for at least 75 days

Exclusion Criteria:

1. Prior or current use of any PPAR-γ agonist
2. Recent use (< 3 months) of an investigational drug
3. Pre-existing medical condition judged to preclude safe participation in the study
4. Contraindication/intolerance to study medication
5. Use of any drug which in the Investigator's opinion could interfere with the glucose level (e.g. systemic corticosteroids)
6. Diagnosed or receiving medication for heart failure, NYHA I to IV
7. Hospitalisation for a major CV event in the last 3 months, scheduled major CV intervention
8. Uncontrolled treated/untreated systolic blood pressure >180 mmHg and/or diastolic blood pressure > 95 mmHg
9. Known diabetic macular oedema
10. Hematuria
11. Serum creatinine >130 μmol/l
12. ALT, AST, total bilirubin or alkaline phosphatase ≥ 2.5 times the upper limit of normal
13. Haemoglobin significantly (in the Investigators opinion, but not more than 1 mmol/L) below the lower limit of normal or haemoglobinopathy interfering with valid HbA1c assay
14. Pregnancy, breast feeding or planning pregnancy or not using adequate contraceptive methods (adequate contraceptive measures are an intrauterine device or oral contraceptives)
15. Mental incapacity, unwillingness, or language barrier precluding adequate understanding or cooperation
16. Abuse of alcohol or drugs, or presence of any condition that in the Investigators opinion may lead to poor adherence to study protocols
17. Cancer or any clinically significant disease or disorder, except for conditions associated to the type 2 diabetes, which in the Investigator's opinion could interfere with the results of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2007-07; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
HbA1c, fasting plasma glucose and 7-point plasma glucose profiles, weight gain, lower leg oedema and safety parameters. | baseline, 4, 8, 12, 17, 21 and 26 weeks

SECONDARY OUTCOMES:
Waist and hip circumferences, plasmaNT-proBNP, ECG, body composition as measured by DXA, blood lipid profiles, plasma insulin | baseline and 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bente J Riis, MD, Study Director — Nordic Bioscience Clinical Studies A/S
Locations (1):
- Multi-center, Copenhagen, Denmark

REFERENCES:
- [Derived] Henriksen K, Byrjalsen I, Qvist P, Beck-Nielsen H, Hansen G, Riis BJ, Perrild H, Svendsen OL, Gram J, Karsdal MA, Christiansen C; BALLET Trial Investigators. Efficacy and safety of the PPARgamma partial agonist balaglitazone compared with pioglitazone and placebo: a phase III, randomized, parallel-group study in patients with type 2 diabetes on stable insulin therapy. Diabetes Metab Res Rev. 2011 May;27(4):392-401. doi: 10.1002/dmrr.1187. PMID 21328517